CLINICAL TRIAL: NCT02597556
Title: A Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Impact of Anthelmintic Treatment on the Incidence of Diarrheal Disease in School Children in Southern Vietnam
Brief Title: The Impact of Anthelmintic Treatment on the Incidence of Diarrheal Disease in Vietnamese School Children
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The prevalence of worm infections in the site is significantly lower than expected
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); Ho Chi Minh Preventive Medicine Centre, Vietnam (Unknown); Princeton University (Other); Cu Chi Health Department (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16EN
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Intestinal Helminthiasis; Diarrhea
Keywords: Albendazole; Ancylostoma duodenale; Ascariasis lumbricoides; Coinfection; Diarrhea; Helminths; Necator americanus; Microbiota; Trichuris trichiura
MeSH Terms: conditions — Intestinal helminthiasis; Diarrhea; Coinfection; Trichuriasis | interventions — Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albendazole (Active Comparator): Albendazole will be administered as a single 400mg chewable tablet at 0, 3, 6, 9, and 12 months.
  Interventions: Drug: Albendazole
- Placebo (Placebo Comparator): Matching Placebo will be administered as a single chewable tablet at 0, 3, 6, and 9 months. At month 12, all participants will receive a single 400mg Albendazole tablet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albendazole — A single 400mg dose of Albendazole administered at 0, 3, 6, 9, and 12 months.
  Arms: Albendazole
Drug: Placebo — Matching placebo tablet administered at 0, 3, 6, and 9 months. At month 12, all participants will receive a single dose of 400mg Albendazole.
  Arms: Placebo

SUMMARY:
Cheap and effective drugs called 'anthelmintics' are routinely administered to children in developing countries to eliminate infections by parasitic helminths. However, the effects of anthelmintic treatment on other pathogens (e.g., bacteria, viruses, protozoa) remain unknown. The aim of this study is to investigate the impact of anthelmintic treatment on the incidence of viral- and bacterial-induced diarrhea in school children in southern Vietnam. Diarrheal disease remains a substantial cause of morbidity and mortality in children in Vietnam, and these children are typically co-infected with intestinal helminths. As helminths and diarrheal pathogens infect the same intestinal niche, anthelmintic treatments may alter host immune responses and the composition of the gut microbiota in ways that affect infection and disease risks caused by diarrheal pathogens.

This study will recruit 350 helminth-infected and 350 helminth-uninfected children aged 6-15 years. Recruited children will be randomized to receive either anthelmintic or placebo treatment once every three months and will be monitored for incidences of diarrheal disease for 12 months. At the 12-month time point, all children will receive anthelmintic treatment. Blood and stool samples will be collected throughout the study and used for evaluation of anemia and host immune responses, and for classification of gut microbes and parasite detection, respectively. The interventional study proposed here will provide an important first test of whether anthelmintic treatments have any indirect effects on infections caused by diarrheal pathogens.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled trial to evaluate the effects of 400 mg albendazole treatment against placebo on the incidence of diarrheal disease caused by viral and bacterial pathogens in school children in southern Vietnam. Children will be enrolled from three primary schools in Cu Chi district in Ho Chi Minh City, Vietnam. Children will be screened for infections by the four most common soil-transmitted helminths, Ascaris lumbricoides, Trichuris trichiura, Necator americanus, and Ancylostoma duodenale. Infected and uninfected individuals will be recruited into the study and randomized to either receive albendazole treatment once every three months for 12 months, or to placebo once every three months for 9 months, after which albendazole treatment will be given at month 12, in accordance with the current deworming schedule in Cu Chi district. A questionnaire regarding the participant's demographics, his/her daily habits, and potential sources of infection will be administered at baseline. Weekly active and passive surveillance of diarrheal cases will be conducted throughout the study, and a health questionnaire will be administered during all cases of diarrhea and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Between 6-15 years of age
* Written informed consent from a parent or guardian
* Written assent from children >10 years of age

Exclusion Criteria:

* Subjects who do not fulfill any component of the inclusion criteria
* Subjects that are both hookworm-positive and anemic, as defined by the WHO guidelines

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of diarrheal disease assessed by 12 months of weekly active and passive case surveillance | 12 months
  Incidence of diarrhea will be defined according to WHO guidelines as three or more loose stools in a 24-hour period or at least one bloody/mucoid stool. To be considered a new episode of diarrhea, at least three intervening days of normal stools without other gastrointestinal symptoms need to have passed between diarrhea occurrences.

SECONDARY OUTCOMES:
Prevalence and intensity of soil-transmitted helminth infections by real-time PCR and microscopy | Baseline, 0.5, 3, 6, 6.5, 9, and 12 months, and during and two weeks after diarrhea cases
Prevalence and intensity of enteric viruses and bacteria that cause diarrhea assessed by real-time PCR and the Luminex xTAG Gastrointestinal Pathogen Panel | Time Frame: Baseline, 3, 6, 9, and 12 months, and during and two weeks after diarrhea cases
Changes in fecal microbiota composition by Illumina sequencing | Baseline, 0.5, 3, 6, 6.5, 9, and 12 months, and during and two weeks after diarrhea cases
Changes in blood cytokine (Th1, Th2, TH17, and Treg) levels by bead-based immunoassays | Baseline, 6, and 12 months of study
Antibody isotype response to helminth and diarrheal antigens by ELISA | Baseline, 6, and 12 months
Mean z-scores (height-for-age, weight-for-age, weight-for-height) | Baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Baker, PhD, Principal Investigator — Oxford University Clinical Research Unit; Nghia Ho Dang Trung, PhD, MD, Principal Investigator — Pham Ngoc Thach University of Medicine; Andrea Graham, PhD, Principal Investigator — Princeton University, USA; Jacqueline Leung, MA, Study Director — Princeton University, USA
Locations (1):
- Cu Chi, Viet Nam, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Blackwell AD, Martin M, Kaplan H, Gurven M. Antagonism between two intestinal parasites in humans: the importance of co-infection for infection risk and recovery dynamics. Proc Biol Sci. 2013 Aug 28;280(1769):20131671. doi: 10.1098/rspb.2013.1671. Print 2013 Oct 22. PMID 23986108
- [Background] Ezenwa VO, Jolles AE. Epidemiology. Opposite effects of anthelmintic treatment on microbial infection at individual versus population scales. Science. 2015 Jan 9;347(6218):175-7. doi: 10.1126/science.1261714. PMID 25574023
- [Background] Ferrari N, Cattadori IM, Rizzoli A, Hudson PJ. Heligmosomoides polygyrus reduces infestation of Ixodes ricinus in free-living yellow-necked mice, Apodemus flavicollis. Parasitology. 2009 Mar;136(3):305-16. doi: 10.1017/S0031182008005404. Epub 2009 Jan 21. PMID 19154651
- [Background] Knowles SC, Fenton A, Petchey OL, Jones TR, Barber R, Pedersen AB. Stability of within-host-parasite communities in a wild mammal system. Proc Biol Sci. 2013 May 15;280(1762):20130598. doi: 10.1098/rspb.2013.0598. Print 2013 Jul 7. PMID 23677343
- [Background] Pedersen AB, Antonovics J. Anthelmintic treatment alters the parasite community in a wild mouse host. Biol Lett. 2013 May 8;9(4):20130205. doi: 10.1098/rsbl.2013.0205. Print 2013 Aug 23. PMID 23658004
- [Background] Nacher M. Worms and malaria: resisting the temptation to generalize. Trends Parasitol. 2006 Aug;22(8):350-1; author reply 351-2. doi: 10.1016/j.pt.2006.06.003. Epub 2006 Jun 23. No abstract available. PMID 16798090
- [Background] Rousham EK. An increase in Giardia duodenalis infection among children receiving periodic Anthelmintic treatment in Bangladesh. J Trop Pediatr. 1994 Dec;40(6):329-33. doi: 10.1093/tropej/40.6.329. PMID 7853436
- [Background] Taylor-Robinson DC, Maayan N, Soares-Weiser K, Donegan S, Garner P. Deworming drugs for soil-transmitted intestinal worms in children: effects on nutritional indicators, haemoglobin, and school performance. Cochrane Database Syst Rev. 2015 Jul 23;2015(7):CD000371. doi: 10.1002/14651858.CD000371.pub6. PMID 26202783
- [Derived] Leung JM, Hong CT, Trung NH, Thi HN, Minh CN, Thi TV, Hong DT, Man DN, Knowles SC, Wolbers M, Hoang Nle T, Thwaites G, Graham AL, Baker S. The impact of albendazole treatment on the incidence of viral- and bacterial-induced diarrhea in school children in southern Vietnam: study protocol for a randomized controlled trial. Trials. 2016 Jun 6;17(1):279. doi: 10.1186/s13063-016-1406-1. PMID 27266697
- See also: Oxford University Clinical research Unit — http://www.oucru.org